CLINICAL TRIAL: NCT06847789
Title: Evaluation of the Tensi+ Device for the Treatment of Overactive Bladder: Prospective Study
Brief Title: Evaluation of the Tensi+ Device for the Treatment of Overactive Bladder
Status: Completed | Type: Observational
Sponsor: Stimuli Technology (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-171221-01 / 1
Record Dates: First submitted 2022-07-08; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Overactive Bladder
Keywords: Urology; TENS; Overactive bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Tensi+ — Tensi+ (Stimuli Technology, Boulogne Billancourt, France) is a newly released, medical transcutaneous-posterior tibial nerve stimulation (TC-pTNS) device marketed for overactive bladder (OAB) management.

SUMMARY:
Tensi+ (Stimuli Technology, Boulogne Billancourt, France) is a newly released, medical transcutaneous-posterior tibial nerve stimulation (TC-pTNS) device marketed for overactive bladder (OAB) management. While effectiveness of TC-pTNS has been demonstrated in the literature, the success rate is heterogeneous, depending on the clinical picture. In an effort to ascertain clearly the efficacy of Tensi+ device, as well as its safety of use and assess comfort of use, the present study will evaluate the results of Tensi+ treatment in real life conditions in a prospective study. The main objective is to assess the efficacy (actual clinical benefit) of TC-pTNS with Tensi+ device for management of overactive bladder in an adult population at 3 months.

Included patients are prescribed a treatment with Tensi+ for 3 months. An evaluation visit is scheduled at 3 months. In treatment is continued, a follow-up visit is scheduled at 6 months.

Primary outcome measure

Success at 3 months defined as a composite parameter:

(i) Objective improvement, with at least 30% decrease of urgency episodes compared to baseline on 3-day bladder diary AND (ii) Subjective improvement, with patient Global Impression of Improvement score of 1 or 2 Time point(s) at which primary outcome measure is assessed : 3 months Secondary outcome measures (i) Evaluation of urinary symptoms based on bladder diary parameters (urinary frequency, incontinence episodes, maximum bladder capacity, nocturia episodes) and the Urinary Symptom Profile (USP) questionnaire (ii) Evaluation of adverse events (iii) Patient-reported Outcomes Measures (PROMs): Comfort of use (VAS in deciles), recommendation to another patient (binary), consumer grading regarding device usability details (iv) Quality of life measures (OABq questionnaire, VAS scale) (vii) Assessment of treatment persistence Time point(s) at which Secondary outcome measure is assessed* : at 3 months and 6 months

Inclusion criteria : Age ≥ 18 years Overactive bladder symptoms

Number of subjects : 100

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients suffering from Overactive bladder symptoms

Exclusion Criteria:

* Pregnancy
* Patients with active implantable device or ankle orthopedic implant,
* Ankle articular diseases.
* Prior treatment with transcutaneous PTNS or percutaneous PTNS (any time),
* Sacral neuromodulation (anytime) or,
* Intradetrusor botulinum toxin injection within the past 6 months
* Antimuscarinic use within 1 month prior to the study
* 24hour diuresis > 2800cc on bladder diary
* Known bladder disease
* Active urinary tract infection
* PVR> 150 ml
* Pelvic organ prolapse stage >2
* Predominant stress urinary incontinence
* Cognitive impairment
* Inability to use the device without a third party
* Inability to complete a bladder diary
* No health insurance coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age ≥ 18 years Overactive bladder symptoms
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Objective improvement | At 3 months
  At least 30% decrease of urgency episodes compared to baseline on 3-day bladder diary
Subjective improvement | At 3 months
  Patient Global Impression of Improvement score of 1 or 2

SECONDARY OUTCOMES:
Evaluation of urinary symptoms | At 3 months and 6 months
  Bladder diary parameters evaluation (urinary frequency, incontinence episodes, maximum bladder capacity, nocturia episodes) and the Urinary Symptom Profile (USP) questionnaire
Evaluation of adverse events | At 3 months and 6 months
  Questions to be asked to patients at 3 months and 6 months if there were any adverse events during treatment
Patient-reported Outcomes Measures (PROMs) | At 3 months and 6 months
  Comfort of use, recommendation to another patient (binary), consumer grading regarding device usability details
Quality of life measures | At 3 months and 6 months
  By filling up OABq questionnaire and VAS scale
Assessment of treatment persistence | At 3 months and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Rouen, Rouen, France

IPD SHARING:
Plan to Share IPD: No